CLINICAL TRIAL: NCT04712812
Title: Registry and Natural History Study for Early Onset Hereditary Spastic Paraplegia (HSP)
Brief Title: Registry and Natural History Study for Early Onset Hereditary Spastic Paraplegia
Acronym: HSP
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Director, Movement Disorders Program, Boston Children's Hospital
Other Study IDs: P00033016
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hereditary Spastic Paraplegia; SPG47; SPG50; SPG51; SPG52; AP4-related Hereditary Spastic Paraplegia; Early Onset Hereditary Spastic Paraplegia; SPG4; SPG3A; SPG15; SPG11
Keywords: AP4-HSP; AP4; SPG; AP-4; AP-4-HSP; Spastic Paraplegia; Adapter Protein 4; HSP; Early onset; Early onset HSP
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Spastic paraplegia 3, autosomal dominant; Paraplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proband with Hereditary Spastic Paraplegia: The study population consists of male and female patients up to the age of 30 years old with a clinical and molecular diagnosis of hereditary spastic paraplegia and/or their family members of interest (if applicable).

SUMMARY:
The Registry and Natural History Study for Early Onset Hereditary Spastic Paraplegia (HSP) is focused on gathering longitudinal clinical data as well as biological samples (skin and/or blood and/or saliva) from male and female patients, under the age of 30, who exhibited early onset symptoms of HSP with (1) a clinical diagnosis of hereditary spastic paraplegia and (2) the presence of variants in HSP related genes and/or be a relative of a person with such a diagnosis. Currently, the treatment for this disorder is generally symptomatic and available therapies improve quality of life, but are grossly inefficient in slowing the disease progression. Access to the registry information will be limited to the study staff who are responsible for recruitment and maintenance of the registry. We hope that recruitment into the registry for studies will advance knowledge of the causes, clinical course, diagnosis, and treatment of these conditions.

DETAILED DESCRIPTION:
The hereditary spastic paraplegias (HSP) are a group of more than 80 neurodegenerative diseases that lead to progressive neurological decline. Collectively, the HSPs present the most common cause of inherited spasticity and associated disability.

We aim to delineate the core clinical, imaging, and molecular features of pediatric onset hereditary spastic paraplegia. This registry and natural history study will facilitate an early diagnosis, enables counseling and anticipatory guidance of affected families and will help define clinically meaningful endpoints for future interventional trials. Samples will be collected for the purpose of molecular and cellular investigation that will help identify biomarkers and novel targets for therapy. The samples and clinical information will be housed in the Translational Neuroscience Center and a secure REDcap database, respectively; both located in Boston Children's Hospital (BCH), but will be available to investigators around the world after approval.

The objectives of this protocol are to (1) To systematically document the clinical presentation and natural history of early-onset forms of HSP and (2) To facilitate an early diagnosis, enable counseling and anticipatory guidance of affected families and help define clinically meaningful endpoints for future interventional traits.

Specifically, the aims are to:

1. Establish the disease spectrum through a cross-sectional analysis of clinical, imaging and molecular data
2. Establish the natural history of early-onset HSP through longitudinal clinician- and patient-reported outcome measures
3. Create a biorepository (blood samples, fibroblasts, induced pluripotent stem cells)
4. Create a registry that allows for re-identification and re-contact of participants by appropriate investigators

ELIGIBILITY:
Inclusion Criteria:

* Onset of hereditary spastic paraplegia symptoms before the age of 18 years
* Under the age of 30 years old
* Must have a genetically confirmed variant in HSP-related genes and a relative of an individual with a confirmed diagnosis (if applicable).

Exclusion Criteria:

* Not having such a diagnosis and/or not being related to such individual

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of male and female patients up to the age of 30 years old with a clinical and molecular diagnosis of hereditary spastic paraplegia and/or their family members of interest (if applicable).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-04-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Establishment of disease spectrum | Through study completion, an average of 1 year
  Establish the disease spectrum through a cross-sectional analysis of clinical, imaging and molecular data
Establishment of longitudinal data | Through study completion, an average of 1 year
  Establish the natural history of early-onset HSP through longitudinal clinician- and patient-reported outcome measures
Creation of biorepository | Through study completion, an average of 1 year
  Create a biorepository (blood samples, fibroblasts, induced pluripotent stem cells)
Creation of patient registry | Through study completion, an average of 1 year
  Create a registry that allows for re-identification and re-contact of participants by appropriate investigators

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Agianda HAP, Kim HM, Battaglia N, Rong J, Tam A, Gonzalez Saez-Diez E, Boerkoel CF, Saffari A, Quiroz V, Schierbaum L, Zaman Z, Bernardi K, Ebrahimi-Fakhari D. Diagnostic Utility of the ATG9A Ratio in AP-4-Associated Hereditary Spastic Paraplegia. Ann Clin Transl Neurol. 2026 Jan 5. doi: 10.1002/acn3.70308. Online ahead of print. PMID 41491634
- [Derived] Schmidt HJD, Battaglia N, Rong J, Tam A, Carty S, Quiroz V, Yang K, Zaman Z, Schierbaum L, Bernardi K, Alecu JE, Ebrahimi-Fakhari D. Health-Related Quality of Life in Rare Forms of Childhood-Onset Hereditary Spastic Paraplegia. Ann Clin Transl Neurol. 2026 Jan;13(1):193-199. doi: 10.1002/acn3.70244. Epub 2025 Nov 6. PMID 41199121